CLINICAL TRIAL: NCT04905394
Title: Short Term Clinical and Radiological Outcomes of Subchondroplasty in the Treatment of Bone Marrow Edema of the Knee
Brief Title: Clinical and Radiological Outcomes of Subchondroplasty in the Treatment of Bone Marrow Edema of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Professor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SubCond
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Bone Marrow Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with subchondroplasty for bone edema in the knee (Experimental): Patients treated with subchondroplasty for bone edema of the knee
  Interventions: Procedure: subchondroplasty

INTERVENTIONS:
Procedure: subchondroplasty — subchondroplasty is an innovative percutaneous procedure in which calcium phosphate, biocompatible material similar to the native bone apatite with osteoinductive properties, is injected inside BML areas. The purpose of subchondroplasty is the patient's symptoms relief, improving the mechanical strength of subchondral bone, stimulating bone remodeling to avoid bone sagging, and slow down the arthritic degenerative process to postpone arthroplasty.

SUMMARY:
Bone marrow lesions (BMLs) of the knee are common subchondral defects, often associated with pain and functional limitation. Subchondroplasty is a percutaneous procedure in which calcium phosphate is injected inside BML areas, ensuring stability and promoting the deposition of new bone. Primary outcome of this study was to obtain a reduction of the Numeric Rating Scale score of 4 points or more at 6 months follow-up in more than 75% of patients. The secondary outcome was to evaluate the osteoarthritic and bone marrow structure evolution in the months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Atraumatic knee pain for at least 3 months;
* Failure of conservative treatment (including NSAIDs, physical therapy, intra- articular injection with steroids or hyaluronic acid and bisphosphonates);
* Mild to moderate osteoarthritis (Kellgren-Lawrence18 grade ≤ 3)
* BML on a loading area at MRI imaging (femoral condyles and/or tibial plateau)

Exclusion Criteria:

* Knee pain and functional limitation related to other causes like osteonecrosis
* Fractures or inflammatory arthritis
* Ligamentous instabilities
* Malalignment on the coronal axis greater than 10 degrees in varus/valgus
* Severe tri-compartmental arthritis (Kellgren-Lawrence grade 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 6 months
  Pain reduction of 4 points in numeric rating score

SECONDARY OUTCOMES:
Radiological evaluation | 6 months
  Evaluation of osteoarthritis progression in the knee on x-rays according to Kellgren&Lawrence classification

CONTACTS AND LOCATIONS:
Overall Officials: pietro randelli, prof, Principal Investigator — University of Milan
Locations (1):
- Gaetano Pini hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Researcher will not share data with other organizations

REFERENCES:
- [Derived] Randelli P, Compagnoni R, Ferrua P, Ricci M, La Verde L, Mekky AF, De Silvestri A, Menon A. Efficacy of Subchondroplasty in the Treatment of Pain Associated With Bone Marrow Lesions in the Osteoarthritic Knee. Orthop J Sports Med. 2023 May 16;11(5):23259671231163528. doi: 10.1177/23259671231163528. eCollection 2023 May. PMID 37213661